CLINICAL TRIAL: NCT01383720
Title: REpositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of Lotus™ Valve SystEm
Acronym: REPRISE I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP3659
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Calcification; Aortic Valve Disease
Keywords: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lotus Valve System (Experimental): Patients enrolled in the study to receive treatment with the Lotus Valve System for symptomatic aortic valve stenosis
  Interventions: Device: Lotus Valve System

INTERVENTIONS:
Device: Lotus Valve System — The Lotus Valve System includes the Lotus Valve, a bovine tissue tri-leaflet bioprosthetic aortic valve, and the Lotus Delivery Catheter for guidance and placement.

SUMMARY:
This is a prospective, single-arm feasibility study designed to assess the acute safety and performance of the Lotus Valve System for transcatheter aortic valve replacement in symptomatic patients with calcified aortic valve stenosis and who are at high risk for surgical intervention.

DETAILED DESCRIPTION:
The incidence of aortic stenosis is increasing due to the aging of the world-wide population and the lack of drug therapies to prevent, halt, or effectively slow the stenotic process. Transcatheter aortic valve replacement has become a viable alternative for treatment of severe symptomatic aortic stenosis in selected patients who are unsuitable candidates for surgical valve replacement. The Lotus Valve System is designed to enable precise placement and minimize or eliminate the paravalvular regurgitation and associated adverse events seen with earlier generation devices. The REPRISE I study assesses acute safety and performance.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 70 years of age or older, and meets all of the criteria below.
2. Patient has documented calcified native aortic valve stenosis, defined with an initial aortic valve area (AVA) of <1.0 cm2 (or AVA index of <0.6 cm2/m2), and a mean pressure gradient >40 mmHg or a jet velocity >4 m/s, as measured by echocardiography.
3. The patient is considered at high risk for surgical aortic valve replacement with an STS (Society of Thoracic Surgeons) score ≥8% or a EuroSCORE ≥20%, or documented multidisciplinary heart team agreement that the patient is at high risk for surgery due to frailty and/or coexisting comorbidities.
4. Symptomatic aortic valve stenosis with New York Heart Association (NYHA) Functional Class ≥ II.
5. Patient has a documented aortic annulus size between 19 and 22 mm (able to accommodate the 23 mm Lotus™ Valve). Pre-procedure measurement by transthoracic echocardiography (TTE) is required. Other imaging modalities (e.g., transesophageal echocardiography (TEE), CT scan) can be used in an adjunctive manner.
6. Patient (or legal representative) understands the trial requirements and the treatment procedures, and provides written informed consent.
7. Patient agrees and is capable of returning to the study hospital for all required scheduled follow up visits.

Exclusion Criteria:

1. Patient has a congenital unicuspid or bicuspid aortic valve.
2. Patient with an acute myocardial infarction (MI) within 30 days of the index procedure (defined as Q wave MI, or non-Q wave MI with total creatine kinase (CK) elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin level elevation (WHO definition)).
3. Patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months, or has any permanent neurologic defect prior to study enrollment.
4. Patient is on dialysis or has serum creatinine level >3.0 mg/dL.
5. Patient has a pre-existing prosthetic heart valve (aortic or mitral) or a prosthetic ring in any position.
6. Patient has >2+ mitral regurgitation or >2+ aortic regurgitation (ie., patient cannot have more than moderate mitral or aortic regurgitation).
7. Moderate to severe pulmonary hypertension (PA systolic pressure >60 mm Hg) as assessed by transthoracic echocardiography.
8. Patient has a need for emergency surgery for any reason.
9. Patient has a history of endocarditis within 12 months of index procedure or evidence of an active systemic infection or sepsis.
10. Patient has echocardiographic evidence of intra-cardiac mass, thrombus or vegetation.
11. Patient has Hgb <9 g/dL, platelet count <100,000 cells/mm3 or >700,000 cells/mm3, and white blood cell (WBC) count <3,000 cells/mm3.
12. Patient is receiving chronic (≥72 hours) anticoagulation therapy (e.g., heparin, warfarin) and who cannot tolerate concomitant therapy with aspirin and clopidogrel (patients who require chronic anticoagulation must be treated with either aspirin or clopidogrel).
13. Patient has active peptic ulcer disease, gastrointestinal (GI) bleed within the past 3 months, other bleeding diathesis or coagulopathy or will refuse transfusions.
14. Patient is contraindicated for transesophageal echocardiography (TEE).
15. Patient has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all thienopyridines, heparin, nickel, titanium, or polyurethanes.
16. Patient has a life expectancy of less than 12 months due to non-cardiac, co-morbid conditions based on the assessment of the investigator at the time of enrollment.
17. Patient has other cardiac devices or hardware with which the study device will interfere with device placement (per physician judgment).
18. Patient has hypertrophic obstructive cardiomyopathy.
19. Patient has any therapeutic invasive cardiac procedure within 30 days prior to the index procedure.
20. Untreated clinically significant coronary artery disease requiring revascularization.
21. Patient has documented left ventricular ejection fraction (LVEF) <30%.
22. Patient is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
23. Patient has severe peripheral vascular disease (including aneurysm defined as maximal luminal diameter >5cm or with documented presence of thrombus, marked tortuosity, narrowing of the abdominal aorta, severe unfolding of the thoracic aorta or thick (>5mm), protruding or ulcerated atheroma in the aortic arch) or symptomatic carotid or vertebral disease.
24. Patient has a femoral artery lumen of <6.0 mm or severe iliofemoral tortuosity or calcification that would prevent safe placement of the introducer sheath.
25. Current problems with substance abuse (e.g. alcohol, cocaine, heroin, etc).
26. Patient is participating in another investigational drug or device study that has not reached its primary endpoint.
27. Patient has preexisting untreated conduction system disorders: Type II second-degree atrioventricular (AV) block, bifascicular or trifascicular block.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Meredith, MBBS, PhD, Principal Investigator — Southern Health, Monash Medical Centre
Locations (3):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St. Vincent's Hospital, Melbourne, Victoria
  - Southern Health Monash Medical Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified by their physicians as meeting the study inclusion/exclusion criteria.
Pre-assignment Details: Screening materials from patients identified by the investigators as having met the inclusion and exclusion criteria were reviewed by a Case Review Committee to assess and confirm eligibility.
Period: Overall Study
Arm/Group | Lotus Valve System
Started | 11
Primary Endpoint (Discharge/7 Days) | 11
Completed | 11 (Study is continuing to 5 years. All patients are still in the study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.0 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Region of Enrollment [Number; unit: participants]
  Australia | 11
General Medical History [Number; unit: participants] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Diabetes mellitus (current) | 5
    Hyperlipidemia (medically treated) | 8
    Hypertension (medically treated) | 10
    History of peripheral vascular disease | 1
    Dialysis dependent renal failure | 0
    Chronic obstructive pulmonary disease | 1
Cardiac History [Number; unit: participants] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Coronary artery disease | 5
    Previous percutaneous coronary intervention | 2
    Previous coronary artery bypass graft surgery | 0
    History of atrial fibrillation | 5
New York Heart Association Class [Number; unit: participants] — New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I (Mild): No limitation of physical activity. Class II (Mild): Slight limitation of physical activity. Class III (Moderate): Marked limitation of physical activity. Class IV (Severe): Unable to carry out any physical activity without discomfort.
  Symptomatic aortic valve stenosis is related to NYHA Functional Class ≥ II.
  participants
    Class I | 0
    Class II | 6
    Class III | 5
    Class IV | 0
Modified Rankin Scale [Number; unit: participants] — Higher score equals a worse condition with zero meaning no symptoms, 2 meaning slight disability and 6 meaning death.
  participants
    0 | 10
    1 | 0
    2 | 1
    3 or higher | 0
Neurological History [Number; unit: participants] — A patient may or may not belong to a category or may belong to more than one category. Therefore the sum may not equal the overall number of patients in the study.
  participants
    Transient Ischemic Attack | 1
    Cerebrovascular Accident | 2
Aortic valve area (effective orifice area) [Mean (Standard Deviation); unit: cm^2] | 0.68 (0.19)
Mean Aortic Valve Gradient [Mean (Standard Deviation); unit: mmHg] | 53.9 (20.9)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percent of LVEF] — This measure represents the percent of Left Ventricular Ejection Fraction.
  percent of LVEF | 62.3 (7.6)
Aortic regurgitation (moderate or severe) [Number; unit: participants] — A patient may or may not belong to a category or may belong to more than one category. Therefore the sum may not equal the overall number of patients in the study.
  participants | 4
Mitral Regurgitation (moderate or severe) [Number; unit: participants] — A patient may or may not belong to a category or may belong to more than one category. Therefore the sum may not equal the overall number of patients in the study.
  participants | 3
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.6 (6.0)
Serum Albumin [Mean (Standard Deviation); unit: g/dL] | 3.9 (0.4)
5-Meter Gait Speed [Mean (Standard Deviation); unit: seconds] | 8.2 (4.9)
Maximum Grip Strength Average [Mean (Standard Deviation); unit: kg] | 15.3 (5.7)
Katz Index [Mean (Standard Deviation); unit: units on a scale] — Katz Index of Independence in Activities of Daily Living (ADL) is an instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently.
  The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
  units on a scale | 5.9 (0.3)
Mini-Cognitive Assessment for Dementia [Mean (Standard Deviation); unit: units on a scale] — Mini-Cognitive Assessment for Dementia scores range from 5 (normal cognition) to 0 (impaired cognition).
  units on a scale | 3.3 (1.5)
Charlson Comorbidity Index Score [Mean (Standard Deviation); unit: units on a scale] — Charlson Comorbidity Index contains 19 categories of comorbidity and assigns a weighted value to each subject's comorbidity based on the risk of 1-year mortality.
  A score of 0 reflects no comorbidities and 19 reveals severe comorbidities.
  units on a scale | 1.8 (1.7)
Society of Thoracic Surgeons (STS) Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons' risk models predict the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. The patient is considered at high risk for surgical aortic valve replacement with an STS score ≥8% or a EuroSCORE ≥20%, or documented multidisciplinary heart team agreement that the patient is at high risk for surgery due to frailty and/or coexisting comorbidities. For example, an STS score of 10% means predicted operative mortality or serious, irreversible morbidity risk of 10% at 30 days.
  units on a scale | 4.9 (2.5)
EuroScore [Mean (Standard Deviation); unit: units on a scale] — European System for Cardiac Operative Risk Evaluation. EuroSCORE is a method of calculating predicted operative mortality for patients undergoing cardiac surgery.
  The patient is considered at high risk for surgical aortic valve replacement with an STS score ≥8% or a EuroSCORE ≥20%, or documented multidisciplinary heart team agreement that the patient is at high risk for surgery due to frailty and/or coexisting comorbidities. EuroScore II is a risk model that calculates the risk of death after a heart operation through 30 days.
  units on a scale | 9.5 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Procedural Success
Description: Clinical procedural success defined as successful implantation of a Lotus Valve System (Device Success) without in-hospital Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) through discharge or 7 days post-procedure, whichever comes first.
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Population: Patients enrolled in the study to receive treatment with the Lotus Valve System for symptomatic aortic valve stenosis
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 9

2. Secondary Outcome: Device Performance Endpoint-Repositioning
Description: Successful repositioning of the Lotus Valve System if repositioning is attempted
Time Frame: procedure
Population: Patients in whom repositioning of the Lotus Valve was attempted
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 4
participants | 4

3. Secondary Outcome: Device Performance Endpoint-Valve Retrieval, if Attempted
Description: Successful retrieval of the Lotus Valve System if retrieval is attempted
Time Frame: procedure
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | NA — There were no attempts made to retrieve the valve.

4. Secondary Outcome: Central Aortic Regurgitation
Description: As determined by echocardiography
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants
  None | 10
  Trivial | 1
  Mild | 0
  Moderate or Severe | 0

5. Secondary Outcome: Paravalvular Aortic Regurgitation
Description: As determined by echocardiography
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants
  None | 8
  Trivial | 1
  Mild | 2
  Moderate or Severe | 0

6. Other Pre Specified Outcome: Successful Access, Device Delivery, Deployment and Positioning and Retrieval of Delivery System
Time Frame: Procedure
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 11

7. Other Pre Specified Outcome: Intended Performance of the Lotus Valve
Description: Aortic valve area >1.0 cm2 plus either a mean aortic valve gradient <20 mmHg or peak velocity <3m/sec, without moderate or severe prosthetic valve aortic regurgitation
Time Frame: At time of discharge or 7 days post procedure
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 10

8. Other Pre Specified Outcome: Single Valve Implanted in the Proper Anatomical Location
Time Frame: procedure
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 11

9. Other Pre Specified Outcome: No Major Adverse Cardiovascular and Cerebrovascular Events Through Discharge
Description: Major adverse cardiovascular or cerebrovascular events include all-cause mortality, periprocedural myocardial infarction ≤72 hours, major stroke, urgent/emergent conversion to surgery or repeat procedure for valve-related dysfunction
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 10

10. Other Pre Specified Outcome: Mean Aortic Valve Gradient
Description: As determined by echocardiography
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
mm Hg | 13.7 (3.7)

11. Other Pre Specified Outcome: Aortic Valve Area
Description: As determined by echocardiography
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
cm^2 | 1.53 (0.18)

12. Other Pre Specified Outcome: Death
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 0

13. Other Pre Specified Outcome: Peri-procedural Myocardial Infarction
Description: Peri-Procedural Myocardial Infarction (≤72 hours after the index procedure)
  * New ischemic symptoms (e.g., chest pain or shortness of breath), or new ischemic signs (e.g. ventricular arrhythmias, new or worsening heart failure, new ST-segment changes, hemodynamic instability, or imaging evidence of new loss of viable myocardium or new wall motion abnormality), AND
  * Elevated cardiac biomarkers (preferably creatine kinase-myoglobin band) within 72 h after the index procedure, consisting of two or more post-procedure samples that are > 0.6 to 8 h apart with a 20% increase in the second sample and a peak value exceeding 10X the 99th percentile upper reference limit (URL), or a peak value exceeding 5X the 99th percentile URL with new pathological Q waves in at least 2 contiguous leads
Time Frame: 72 hours
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 0

14. Other Pre Specified Outcome: Major Stroke
Description: Confirmed with a Modified Rankin score >/= 2 at 30 and 90 days
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 1

15. Other Pre Specified Outcome: Urgent/Emergent Conversion to Surgery or Repeat Procedure for Valve-related Dysfunction
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 0

16. Other Pre Specified Outcome: Major Vascular Complication
Description: * Any thoracic aortic dissection
  * Access site or access-related vascular injury (dissection, stenosis, perforation, rupture, arterio-venous fistula, pseudoaneurysm, hematoma, irreversible nerve injury, or compartment syndrome) leading to either death, need for significant blood transfusions (≥4 units), unplanned percutaneous or surgical intervention, or irreversible end-organ damage (e.g. hypogastric artery occlusion causing visceral ischemia or spinal artery injury causing neurologic impairment)
  * Distal embolization (non-cerebral) from a vascular source requiring surgery or resulting in amputation or irreversible end-organ damage
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 1

17. Other Pre Specified Outcome: New Conduction Disturbances or Arrhythmias Requiring Permanent Pacemaker
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 4

18. Other Pre Specified Outcome: Bleeding
Description: Life-threatening or Disabling Bleeding
  * Fatal bleeding OR
  * Bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome OR
  * Bleeding causing hypovolemic shock or severe hypotension requiring vasopressors or surgery OR
  * Overt source of bleeding with drop in hemoglobin of ≥5 g/dL or whole blood or packed red blood cells (RBC) transfusion ≥4 units
  Major Bleeding
  * Overt bleeding either associated with a drop in the hemoglobin level of at least 3.0g/dL or requiring transfusion of 2 or 3 units of whole blood/RBC AND
  * Does not meet criteria of life-threatening or disabling bleeding
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants
  Life-threatening or disabling | 0
  Major | 2

19. Other Pre Specified Outcome: Acute Kidney Injury - Stage 2 or 3
Description: Stage 2: Increase in serum creatinine to 200-300% (2.0-3.0 times increase compared with baseline).
  Stage 3: Increase in serum creatinine to ≥ 300% (> 3 times increase compared with baseline) or serum creatinine of ≥ 4.0 mg/d (≥ 354 μmol/L) with an acute increase of at least 0.5 mg/dl (44 μmol/L). Subjects receiving renal replacement therapy are considered to meet Stage 3 criteria irrespective of other criteria.
Time Frame: Discharge or 7 days post-procedure, whichever comes first
Measure: Number; unit: participants
Arm/Group | Lotus Valve System
Number analyzed (Participants) | 11
participants | 0

ADVERSE EVENTS:
Time Frame: After 1 year index procedure
Arm/Group | Lotus Valve System
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotus Valve System (N=11)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotus Valve System (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 7 (7)
Myocardial infarction (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Secretion discharge (General disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 3 (3)
Peripheral artery dissection (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to the Sponsor for review at least 45 days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.